CLINICAL TRIAL: NCT00149214
Title: A Randomized Phase 2 Trial of Doxorubicin Plus Pemetrexed Followed by Docetaxel, Versus Doxorubicin Plus Cyclophosphamide Followed by Docetaxel, as Neoadjuvant Treatment for Early Breast Cancer
Brief Title: Preoperative Treatment of Breast Cancer With Two Different Sequential Treatment Regimens
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7113; H3E-MC-S080 (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-02; First posted 2005-09-08 (Estimated); Results first posted 2009-05-13 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Pemetrexed; Cyclophosphamide; Doxorubicin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Pemetrexed Plus Doxorubicin, Followed by Docetaxel (Experimental)
  Interventions: Drug: pemetrexed; Drug: doxorubicin; Drug: docetaxel
- B: Cyclophosphamide Plus Doxorubicin, Followed by Docetaxel (Active Comparator)
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin; Drug: docetaxel

INTERVENTIONS:
Drug: pemetrexed — 500 mg/m^2, intravenous (IV), every 21 days, 4 cycles (1-4)
  Other Names: LY231514, Alimta
  Arms: A: Pemetrexed Plus Doxorubicin, Followed by Docetaxel
Drug: cyclophosphamide — 600 mg/m2, intravenous (IV), every 21 days, 4 cycles (1-4)
  Arms: B: Cyclophosphamide Plus Doxorubicin, Followed by Docetaxel
Drug: doxorubicin — 60 mg/m^2, intravenous (IV), every 21 days, 4 cycles (1-4)
Drug: docetaxel — 100 mg/m^2, intravenous (IV), every 21 days, 4 cycles (5-8)

SUMMARY:
An open-label randomized Phase II study in order to explore two different sequential anthracycline-based neoadjuvant treatment regimens in female patients with primary, operable breast cancer (T2-T4/N0-2/M0).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of primary early breast cancer, tumor size greater than or equal to 2 centimeters (cm), of Stages T2-T4/N0-2.
* Performance status 0-2 Eastern Cooperative Oncology Group (ECOG).
* Adequate organ function (bone marrow, hepatic, renal, cardiac).

Exclusion Criteria:

* Prior anthracyclines as part of prior anticancer therapy.
* Concurrent antitumor therapy.
* Second primary malignancy.
* Serious concomitant systemic disorder.
* Pre-existing sensorial or motor neuropathy

  * Grade 1.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2005-09; Primary Completion 2008-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Monday-Friday 9am - 5pm Eastern time (UTC/GMT - 5 hours, EST), Study Chair — Eli Lilly and Company
Locations (11):
- Germany (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baden-Baden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
- Italy (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cremona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rozzano
- Russia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
- Spain (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jaén
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sabadell
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia

REFERENCES:
- [Result] Schneeweiss A, Marme F, Ruiz A, Manikhas AG, Bottini A, Wolf M, Sinn HP, Mansouri K, Kennedy L, Bauknecht T. A randomized phase II trial of doxorubicin plus pemetrexed followed by docetaxel versus doxorubicin plus cyclophosphamide followed by docetaxel as neoadjuvant treatment of early breast cancer. Ann Oncol. 2011 Mar;22(3):609-617. doi: 10.1093/annonc/mdq400. Epub 2010 Aug 23. PMID 20732932
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The one participant who was randomized to pemetrexed but treated with cyclophosphamide is included in the as randomized group (pemetrexed) for the purposes of the participant flow, excluded from the efficacy analyses (per the protocol), but in the as treated group (cyclophosphamide) for safety analyses.
Groups:
- Pemetrexed Plus Doxorubicin, Followed by Docetaxel: pemetrexed: 500 mg/m^2, intravenous (IV), every 21 days, 4 cycles (1-4) doxorubicin: 60 mg/m^2, intravenous (IV), every 21 days, 4 cycles (1-4) docetaxel: 100 mg/m^2, intravenous (IV), every 21 days, 4 cycles (5-8)
- Cyclophosphamide Plus Doxorubicin, Followed by Docetaxel: cyclophosphamide: 600 mg/m^2, intravenous (IV), every 21 days, 4 cycles (1-4) doxorubicin: 60 mg/m^2, intravenous (IV), every 21 days, 4 cycles (1-4) docetaxel: 100 mg/m^2, intravenous (IV), every 21 days, 4 cycles (5-8)
Period: Overall Study
Arm/Group | Pemetrexed Plus Doxorubicin, Followed by Docetaxel | Cyclophosphamide Plus Doxorubicin, Followed by Docetaxel
Started | 135 (One patient randomized to Pemetrexed (P) was treated with Cyclophosphamide (C).) | 122
Completed | 109 (The patient treated with Cyclophosphamide (C) was included in that arm (C) for safety analysis.) | 105
Not Completed | 26 | 17
Not completed — Adverse Event | 12 | 9
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Physician Decision | 3 | 3
Not completed — Sponsor Decision | 0 | 1
Not completed — Progressive Disease | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed Plus Doxorubicin, Followed by Docetaxel | Cyclophosphamide Plus Doxorubicin, Followed by Docetaxel | Total
Number analyzed (Participants) | 135 | 122 | 257
Age Continuous [Mean (Standard Deviation); unit: years] | 49.9 (10.2) | 49.5 (9.7) | 49.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 122 | 257
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 36 | 29 | 65
  Russian Federation | 14 | 14 | 28
  Germany | 74 | 71 | 145
  Italy | 11 | 8 | 19
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants]
  Grade 0 - Fully active | 131 | 113 | 244
  Grade 1- Ambulatory; strenuous activity restricted | 1 | 4 | 5
  Status Unknown | 3 | 5 | 8
Estrogen and Progesterone Receptor Status [Number; unit: participants]
  At least one positive | 90 | 78 | 168
  Both negative | 45 | 44 | 89
Menopausal Status [Number; unit: participants]
  Unknown | 0 | 1 | 1
  Pre-Menopausal | 69 | 66 | 135
  Peri-Menopausal | 6 | 7 | 13
  Post-Menopausal | 60 | 48 | 108
Race/Ethnicity [Number; unit: participants]
  Caucasian | 135 | 119 | 254
  Hispanic | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Pathological Complete Response
Description: pathological assessment of tissue removed during surgery to determine if tumor tissue is still present after chemotherapy
Time Frame: surgery after eight 21-day cycles of chemotherapy
Population: Participants meeting the following criteria qualify for pathological tumor response:
  * Histologic diagnosis of primary operable breast cancer
  * No concurrent antitumor therapy
  * Specimen for evaluation of pathological response obtained upon surgery
  * Treatment with at least one dose of study drug of the assigned study regimen.
Measure: Number; unit: participants
Arm/Group | Pemetrexed Plus Doxorubicin, Followed by Docetaxel | Cyclophosphamide Plus Doxorubicin, Followed by Docetaxel
Number analyzed (Participants) | 127 | 119
participants
  Pathological Complete Response | 21 | 24
  Tumor Cells Still Present | 99 | 89
  Not evaluable | 7 | 6
Statistical Analysis 1: Comparison: Pemetrexed Plus Doxorubicin, Followed by Docetaxel; Confidence Interval for pathological complete response in the Pemetrexed treatment arm; Test type: Superiority or Other; Percentage of Participants = 16.5, 95% CI [10.5 to 24.2]
Statistical Analysis 2: Comparison: Cyclophosphamide Plus Doxorubicin, Followed by Docetaxel; Confidence Interval for pathological complete response in the Cyclophosphamide treatment group; Test type: Superiority or Other; Percentage of Participants = 20.2, 95% CI [13.4 to 28.5]

2. Secondary Outcome: Number of Participants With a Clinical Tumor Response After the First Sequence of Chemotherapy
Description: The number of participants with a clinical tumor response based on measurement of tumor size after the first sequence of chemotherapy, without a second confirmatory tumor measurement, per protocol.
Time Frame: Cycles 1-4 (21-day cycles)
Population: Participants meeting following criteria qualify for clinical tumor response:
  * Histologic diagnosis of primary operable breast cancer
  * No concurrent antitumor therapy up to surgery
  * Presence of measurable disease as defined by RECIST.
  * Treatment with at least one dose of study drug of assigned study regimen.
Measure: Number; unit: participants
Arm/Group | Pemetrexed Plus Doxorubicin, Followed by Docetaxel | Cyclophosphamide Plus Doxorubicin, Followed by Docetaxel
Number analyzed (Participants) | 131 | 119
participants
  Complete Response | 8 | 9
  Partial Response | 45 | 43
  Stable Disease | 49 | 44
  Progressive Disease | 3 | 2
  Unknown | 17 | 17
  Not Done | 9 | 4

3. Secondary Outcome: Number of Participants With a Clinical Tumor Response After the Second Sequence of Chemotherapy
Description: The number of participants with a clinical tumor response based on measurement of tumor size after the second sequence of chemotherapy, without a second confirmatory tumor measurement required, per protocol.
Time Frame: Cycles 5-8 (21-day cycles)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Pemetrexed Plus Doxorubicin, Followed by Docetaxel | Cyclophosphamide Plus Doxorubicin, Followed by Docetaxel
Number analyzed (Participants) | 131 | 119
participants
  Complete Tumor Response | 19 | 21
  Partial Tumor Response | 59 | 60
  Stable Disease | 35 | 24
  Progressive Disease | 2 | 1
  Unknown | 9 | 10
  Not Done | 7 | 3

4. Secondary Outcome: Number of Patients With Histologically Negative Axillary Lymph Node Status at Surgery
Description: Histologically negative is defined as no malignant cells present in the axillary lymph nodes during surgery.
Time Frame: surgery after eight 21-day cycles of chemotherapy
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Pemetrexed Plus Doxorubicin, Followed by Docetaxel | Cyclophosphamide Plus Doxorubicin, Followed by Docetaxel
Number analyzed (Participants) | 127 | 119
participants | 64 | 63

5. Secondary Outcome: Disease-free Survival
Description: Disease-free survival is defined as the time from date of study enrollment (randomization) to first date of progressive disease (PD) or death from any cause. PD per Response Evaluation Criteria In Solid Tumors (RECIST) criteria is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. For patients not known to have died as of the data cut-off date and who do not have progressive disease, disease-free survival was censored at the last contact date.
Time Frame: baseline through post surgery, follow-up for 3 years post-surgery (up to 5.2 years after randomization)
Population: All randomized participants. In the Pemetrexed plus Doxorubicin, Followed by Docetaxel arm, 99 participants were censored. In the Cyclophosphamide plus Doxorubicin, Followed by Docetaxel arm, 94 participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed Plus Doxorubicin, Followed by Docetaxel | Cyclophosphamide Plus Doxorubicin, Followed by Docetaxel
Number analyzed (Participants) | 135 | 122
months | NA [47.96 to NA] — The median and upper limit of the 95% confidence interval were not calculable because an insufficient number of participants reached the event at the final time point for assessment. | NA [54.38 to NA] — The median and upper limit of the 95% confidence interval were not calculable because an insufficient number of participants reached the event at the final time point for assessment.

ADVERSE EVENTS:
Arm/Group | Pemetrexed Plus Doxorubicin, Followed by Docetaxel | Cyclophosphamide Plus Doxorubicin, Followed by Docetaxel
Serious Adverse Events (participants affected / at risk) | 15/134 | 25/123
Other Adverse Events (participants affected / at risk) | 134/134 | 120/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed Plus Doxorubicin, Followed by Docetaxel (N=134) | Cyclophosphamide Plus Doxorubicin, Followed by Docetaxel (N=123)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5) | 5 (6)
Leukopenia (Blood and lymphatic system disorders) | 4 (4) | 9 (9)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1)
Injection site extravasation (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 5 (5)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia primary atypical (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Vulvitis (Infections and infestations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Axillary vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Post procedural haematoma (Vascular disorders) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed Plus Doxorubicin, Followed by Docetaxel (N=134) | Cyclophosphamide Plus Doxorubicin, Followed by Docetaxel (N=123)
Anaemia (Blood and lymphatic system disorders) | 10 (17) | 11 (19)
Leukocytosis (Blood and lymphatic system disorders) | 13 (29) | 9 (18)
Leukopenia (Blood and lymphatic system disorders) | 66 (229) | 67 (252)
Lymphopenia (Blood and lymphatic system disorders) | 19 (53) | 18 (50)
Neutropenia (Blood and lymphatic system disorders) | 65 (223) | 73 (244)
Neutrophilia (Blood and lymphatic system disorders) | 7 (14) | 4 (7)
Thrombocythaemia (Blood and lymphatic system disorders) | 9 (12) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (18) | 12 (22)
Conjunctivitis (Eye disorders) | 19 (32) | 10 (14)
Lacrimation increased (Eye disorders) | 16 (20) | 14 (15)
Abdominal pain (Gastrointestinal disorders) | 16 (18) | 12 (17)
Abdominal pain upper (Gastrointestinal disorders) | 21 (24) | 11 (12)
Constipation (Gastrointestinal disorders) | 49 (81) | 35 (51)
Diarrhoea (Gastrointestinal disorders) | 33 (50) | 27 (42)
Dyspepsia (Gastrointestinal disorders) | 10 (11) | 9 (9)
Nausea (Gastrointestinal disorders) | 82 (207) | 81 (210)
Stomatitis (Gastrointestinal disorders) | 53 (95) | 47 (90)
Vomiting (Gastrointestinal disorders) | 30 (43) | 40 (69)
Asthenia (General disorders) | 34 (90) | 28 (75)
Chills (General disorders) | 9 (9) | 11 (11)
Fatigue (General disorders) | 49 (100) | 45 (106)
Mucosal inflammation (General disorders) | 27 (47) | 18 (24)
Pain (General disorders) | 8 (9) | 8 (8)
Pyrexia (General disorders) | 21 (30) | 21 (28)
Nasopharyngitis (Infections and infestations) | 6 (6) | 9 (9)
Alanine aminotransferase (Investigations) | 22 (30) | 7 (10)
Alanine aminotransferase increased (Investigations) | 57 (87) | 33 (40)
Aspartate aminotransferase (Investigations) | 22 (29) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 54 (80) | 29 (32)
Blood alkaline phosphatase increased (Investigations) | 5 (5) | 7 (11)
Blood glucose increased (Investigations) | 11 (25) | 6 (13)
Blood lactate dehydrogenase increased (Investigations) | 26 (33) | 15 (23)
Gamma-glutamyltransferase increased (Investigations) | 8 (11) | 7 (8)
Haemoglobin (Investigations) | 9 (11) | 6 (7)
Haemoglobin decreased (Investigations) | 32 (83) | 38 (86)
Neutrophil count (Investigations) | 9 (21) | 4 (9)
Neutrophil count decreased (Investigations) | 15 (38) | 9 (21)
Neutrophil count increased (Investigations) | 10 (22) | 12 (23)
Platelet count increased (Investigations) | 8 (11) | 5 (6)
Red blood cell count decreased (Investigations) | 7 (9) | 4 (7)
White blood cell count (Investigations) | 10 (18) | 6 (15)
White blood cell count decreased (Investigations) | 13 (28) | 8 (19)
White blood cell count increased (Investigations) | 12 (23) | 12 (22)
Anorexia (Metabolism and nutrition disorders) | 22 (34) | 25 (47)
Fluid retention (Metabolism and nutrition disorders) | 20 (23) | 14 (16)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (21) | 8 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 (56) | 28 (59)
Bone pain (Musculoskeletal and connective tissue disorders) | 16 (16) | 16 (21)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 (14) | 10 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (23) | 21 (30)
Dizziness (Nervous system disorders) | 6 (9) | 8 (9)
Dysgeusia (Nervous system disorders) | 20 (27) | 26 (37)
Headache (Nervous system disorders) | 12 (14) | 20 (26)
Peripheral sensory neuropathy (Nervous system disorders) | 15 (25) | 12 (18)
Polyneuropathy (Nervous system disorders) | 25 (32) | 24 (31)
Insomnia (Psychiatric disorders) | 7 (9) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 12 (14)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 80 (88) | 68 (75)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (8) | 9 (10)
Erythema (Skin and subcutaneous tissue disorders) | 19 (31) | 17 (29)
Nail disorder (Skin and subcutaneous tissue disorders) | 38 (47) | 35 (45)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 14 (17) | 13 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (11) | 14 (16)
Rash (Skin and subcutaneous tissue disorders) | 14 (14) | 4 (6)
Hot flush (Vascular disorders) | 6 (7) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days